CLINICAL TRIAL: NCT06744114
Title: Etiologies, Definitive Diagnosis and Patient Outcomes in Altered Level of Consciousness in the Emergency Department
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHS/Batch-Spring23/017
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Consciousness Disorders
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Consciousness in the Emergency Department — To determine the common and definitive etiologies of altered level of consciousness in emergency department.

SUMMARY:
When someone starts acting differently in terms of how alert or awake they are, it can be a tough situation for emergency (ER) department doctors.e exact and definitive etiologies of ALOC that can be intracranial or extracranial.

DETAILED DESCRIPTION:
The change in terms of mental state in accordance with how alert and awake patient is termed as altered level of consciousness. Etiologies will be classified by using convenience sampling. GCS<14 patients will be included in this study. Data will be collected through a slight modification in a pre-designed Performa. Reference point for the data collection will be the time of discharge from the emergency department. In Previous studies mostly, etiologies were classified as extracranial and intracranial. Some studies found neurological etiologies most dominant as an extra cranial and some studies found systematic infections ,metabolic causes and some demonstrated that intracranial etiologies were dominant. So, in this study we will find the definitive diagnosis in patient having ALOC which can be intracranial or extracranial. And also, it will be compared with GCS scale. This study will identify th

ELIGIBILITY:
Inclusion Criteria:

* Patients with GCS<15, age group 18 years to 90 years which come in emergency department due to any etiology will be included in this study.

Exclusion Criteria:

* GCS = 15 will be excluded from the study.
* patients coming in any outpatient department setting or other than emergency department and age group <18 or > 90 will be excluded from this study.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Definitive Diagnosis and Patient Outcomes in Altered Level of Consciousness in the Emergency Department
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
GCS(GLASGOW COMMA SCALE) | 12 Months
  The GCS is scored between 3 and 15, 3 being the worst and 15 the best. It is composed of three parameters: best eye response (E), best verbal response (V), and best motor response (M). The components of the GCS should be recorded individually.

CONTACTS AND LOCATIONS:
Locations (1):
- CMH RAWALAKOT AJK, District poonch , tehsil Rawalakot, AJK PAKISTAN, Kashmir, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No